CLINICAL TRIAL: NCT07169448
Title: Impact of A Postoperative Meal Delivery Program on Malnutrition in Orthopaedic Trauma Patients
Brief Title: Food is Medicine Prospective Study
Acronym: FIM
Status: Not yet recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Carol A. Lin, MD, Associate Professor, Cedars-Sinai Medical Center
Other Study IDs: STUDY00004008
Record Dates: First submitted 2025-08-25; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Wounds and Injuries
Keywords: Food is medicine
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopaedic trauma surgical patients with inpatient stay: Discharged home from hospital, skilled nursing facility, or acute rehab

SUMMARY:
The purpose of this study is to examine the impact of a medically tailored post-operative meal delivery program on surgical outcomes and metabolic lab markers in orthopaedic trauma patients. Patients will have 12 days of meals and shakes delivered to their house through our partnership with Meals on Wheels. Metabolic lab values will be drawn at the 2 week and 6 week post-op visits. All patients will be followed for up to 1 year postoperatively.

DETAILED DESCRIPTION:
This project addresses critical gaps in our understanding of how malnutrition affects recovery in orthopaedic trauma patients by focusing on three key outcomes: (1) the incidence of acute wound complications, (2) metabolic biomarker changes over time, and (3) patient-reported outcomes (PROMIS scores) and impact (qualitative survey) during the recovery period. By systematically investigating these outcomes, the project aims to understand how post-operative meal supplementation can be optimized to reduce complications and improve recovery. The findings will have significant implications for clinical practice, particularly in developing nutritional programs and guidelines that can be integrated into post-operative care protocols to improve outcomes and reduce healthcare costs for orthopaedic trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years old or older are included.
* English or Spanish speaking
* Reside in the following zip codes: 90001, 90002, 90003, 90004, 90005, 90006, 90007, 90008, 90009, 90010, 90011, 90012, 90013, 90014, 90015, 90016, 90017, 90018, 90019, 90020, 90021, 90023, 90026, 90027, 90028, 90029, 90031, 90035, 90036, 90037, 90038, 90039, 90043, 90044, 90046, 90047, 90048, 90052, 90057, 90059, 90061, 90062, 90065, 90068, 90069
* Discharged home, either directly from Cedars-Sinai Medical Center or after time in a skilled nursing facility or acute rehab
* Orthopaedic trauma surgical patients that have had an operation and inpatient stay at Cedars-Sinai Medical Center

Exclusion Criteria:

* Any records flagged "break the glass" or "research opt out."
* Any pregnant patients.
* Patients with any congenital metabolic conditions
* Patients with dietary restrictions (ex. Kosher, Halal, vegan, gluten free, etc.) that are unable to be reasonably accommodated by St. Vincent Meals on Wheels
* Any patients with mental illness the prevents them from giving consent.
* Patients with dementia or cognitive impairment.
* Patients who are homeless and/or unreliable to follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic trauma surgical patients that have had an operation and inpatient stay at Cedars-Sinai Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Metabolic biomarker changes over time | From enrollment to 6-weeks postop
  Evaluation of biomarkers
Incidence of acute wound complications | From enrollment to end of treatment at 1-year postop
  Wound compliaction

OTHER OUTCOMES:
Patient-reported outcomes Depression | From enrollment to end of study period at 1-year postop
  The PROMIS Depression scale is a self-reported measure used to assess negative mood, views of self, and social cognition associated with depressive symptoms. Scores are reported on a T-score metric, standardized with a mean of 50 and standard deviation of 10, based on the U.S. general population.
  Scale Range: 0 to 100 (T-score)
  Interpretation: Higher scores indicate worse outcomes, meaning more severe depressive symptoms.
  A T-score of 50 represents the average level of depressive symptoms in the general population.
Patient-reported outcomes Anxiety | From enrollment to end of study period at 1-year postop
  The PROMIS Anxiety scale measures fear, anxious misery, hyperarousal, and somatic symptoms related to anxiety. Like other PROMIS instruments, it uses a T-score metric with a mean of 50 and standard deviation of 10.
  Scale Range: 0 to 100 (T-score)
  Interpretation: Higher scores indicate worse outcomes, meaning greater severity of anxiety symptoms.
  A T-score of 50 reflects the average level of anxiety symptoms in the general population.
Patient-reported outcomes Physical Function | From enrollment to end of study period at 1-year postop
  The PROMIS Physical Function scale evaluates an individual's capability to perform physical activities such as mobility, dexterity, and self-care. Scores are reported using a T-score, standardized with a mean of 50 and standard deviation of 10.
  Scale Range: 0 to 100 (T-score)
  Interpretation: Higher scores indicate better outcomes, meaning greater physical functioning.
  A T-score of 50 reflects the average physical function in the general population.
Patient-reported outcomes Pain Interference | From enrollment to end of study period at 1-year postop
  The PROMIS Pain Interference scale assesses the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. It is scored on the T-score metric, with a mean of 50 and standard deviation of 10.
  Scale Range: 0 to 100 (T-score)
  Interpretation: Higher scores indicate worse outcomes, meaning pain is interfering more with daily life.
  A T-score of 50 indicates average pain interference relative to the general population.

CONTACTS AND LOCATIONS:
Overall Officials: Milton Little, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Firoozabadi R, Hamilton B, O'Donnell C, Agel J, Benirschke S, Kramer P, Henley MB. Prospective Study Investigating the Prevalence and Evolution of Malnourishment in the Acute Orthopaedic Trauma Patient. Arch Bone Jt Surg. 2022 Jul;10(7):592-600. doi: 10.22038/ABJS.2021.47718.2341. PMID 36032641
- [Background] George A, Holderread BM, Lambert BS, Harris JD, McCulloch PC. Post-operative protein supplementation following orthopaedic surgery: A systematic review. Sports Med Health Sci. 2023 Sep 7;6(1):16-24. doi: 10.1016/j.smhs.2023.08.002. eCollection 2024 Mar. PMID 38463662
- [Background] Lawson RM, Doshi MK, Barton JR, Cobden I. The effect of unselected post-operative nutritional supplementation on nutritional status and clinical outcome of orthopaedic patients. Clin Nutr. 2003 Feb;22(1):39-46. doi: 10.1054/clnu.2002.0588. PMID 12553948
- [Background] Yeung SE, Hilkewich L, Gillis C, Heine JA, Fenton TR. Protein intakes are associated with reduced length of stay: a comparison between Enhanced Recovery After Surgery (ERAS) and conventional care after elective colorectal surgery. Am J Clin Nutr. 2017 Jul;106(1):44-51. doi: 10.3945/ajcn.116.148619. Epub 2017 May 3. PMID 28468890
- [Background] Mosquera C, Koutlas NJ, Edwards KC, Strickland A, Vohra NA, Zervos EE, Fitzgerald TL. Impact of malnutrition on gastrointestinal surgical patients. J Surg Res. 2016 Sep;205(1):95-101. doi: 10.1016/j.jss.2016.05.030. Epub 2016 May 26. PMID 27621004
- [Background] Handcox JE, Gutierrez-Naranjo JM, Salazar LM, Bullock TS, Griffin LP, Zelle BA. Nutrition and Vitamin Deficiencies Are Common in Orthopaedic Trauma Patients. J Clin Med. 2021 Oct 28;10(21):5012. doi: 10.3390/jcm10215012. PMID 34768533
- [Background] Ernst A, Wilson JM, Ahn J, Shapiro M, Schenker ML. Malnutrition and the Orthopaedic Trauma Patient: A Systematic Review of the Literature. J Orthop Trauma. 2018 Oct;32(10):491-499. doi: 10.1097/BOT.0000000000001254. PMID 30247276
- [Background] Leandro-Merhi VA, de Aquino JL. Determinants of malnutrition and post-operative complications in hospitalized surgical patients. J Health Popul Nutr. 2014 Sep;32(3):400-10. PMID 25395903
- [Background] Bonilla-Palomas JL, Gamez-Lopez AL, Castillo-Dominguez JC, Moreno-Conde M, Lopez Ibanez MC, Alhambra Exposito R, Ramiro Ortega E, Anguita-Sanchez MP, Villar-Raez A. Nutritional Intervention in Malnourished Hospitalized Patients with Heart Failure. Arch Med Res. 2016 Oct;47(7):535-540. doi: 10.1016/j.arcmed.2016.11.005. PMID 28262195
- [Background] Ponsford J, Hill B, Karamitsios M, Bahar-Fuchs A. Factors influencing outcome after orthopedic trauma. J Trauma. 2008 Apr;64(4):1001-9. doi: 10.1097/TA.0b013e31809fec16. PMID 18404068
- [Background] Kehlet H, Wilmore DW. Multimodal strategies to improve surgical outcome. Am J Surg. 2002 Jun;183(6):630-41. doi: 10.1016/s0002-9610(02)00866-8. PMID 12095591